CLINICAL TRIAL: NCT04911205
Title: Efficacy of High Intensity Preoperative Training on Postoperative Outcomes in Greek Patients Undergoing Total Knee Arthroplasty: a Randomized Controlled Study
Brief Title: Preoperative Rehabilitation in Greek Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Dimitrios Vasileiadis, Principal Investigator Mr Dimitrios Vasileiadis, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1819019724
Record Dates: First submitted 2021-05-26; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis; Rehabilitation
Keywords: physiotherapy; preoperative rehabilitation; osteoarthritis; total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients who were randomly allocated to intervention group (N=44) completed a 6-week preoperative training program, 5 days per week prior to surgery
  Interventions: Other: Preoperative training program
- Control Group (No Intervention): Patients who were randomly allocated to control group (N=44), they continued to live as usual, prior to surgery

INTERVENTIONS:
Other: Preoperative training program — Patients of intervention group (N=44) followed a 6-week supervised high-intensity preoperative training program. They had a session of preoperative resistance training five days per week for a period of 6 weeks before TKA. Each session was supervised by a physiotherapist specifically trained in progressive resistance training. The duration of each session was approximately 60 minutes. If a participant missed a training session, it was attempted to substitute the session on an alternative day.
  Arms: Intervention Group

SUMMARY:
Purpose: The purpose of this study was to investigate the efficacy of a 6-week supervised high-intensity preoperative training program on muscle strength, functional performance and patient-reported outcomes in patients undergoing total knee arthroplasty (TKA).

Methods: Eighty-eight patients scheduled for unilateral TKA for severe osteoarthritis (OA) were randomly allocated to intervention group (N=44) completed a 6-week preoperative training program, 5 days per week prior to surgery and to control group (N=44) who lived as usual. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), the Physical Functioning Scale of the Short Form-36 questionnaire (SF-36), Knee Injury and Osteoarthritis Outcome Score (KOOS), quadriceps strength, 20 meters walk test and 30 seconds chair stand test were assessed at 6 weeks before surgery (T0), after 6 weeks of preoperative training / preoperatively (T1), 4 weeks (T2) and finally 12 weeks (T3) after TKA.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the efficacy of 6 weeks of preoperative and 4-week postoperative progressive resistance training (PRT) compared to 4 weeks of postoperative PRT only on functional performance, muscle strength, and patient-reported outcomes in patients undergoing TKA. We hypothesized that 6 weeks of preoperative PRT would be safe and feasible and would improve functional performance, knee extensor and flexor muscle strength, and patient-reported outcomes preoperatively and at 4 and 12 weeks postoperatively, when compared to controls.

Materials and methods

All patients over 60 years old who were diagnosed with advanced idiopathic knee OA (according to the radiological criteria of the American College of Rheumatology Guidelines) and scheduled for unilateral total knee arthroplasty in Orthopedic Clinic of University Hospital of Alexandroupolis, Greece from March 2014 until January 2016 were considered candidates for this study and were informed to participate. Exclusion criteria were medical conditions that exercise was contraindicated (i.e cardiopulmonary comorbidities that precluded modest exercise), diseases that affected their functional performance (suffering from neuromuscular or neurodegenerative conditions), mental diseases, previous hip or knee joint replacement surgery and if they had severe pain in the controlateral limp that would not allow them to follow any pre- or postoperative interventions.

Eligible participants signed an informed consent document approved by The Research Ethics Committee of the Faculty of Health Sciences, National and Kapodistrian University of Athens,(16955 : 03/12/2018) prior to participation in the study. This study took a clinical trial number (registration number 1819019724/23-01-2019) from National and Kapodistrian University of Athens, Greece.

Of the total 234 patients screened, 88 patients were finally included to our study and 136 were excluded. O those, 85 declined to participate and 51 did not meet the inclusion criteria. Patients (N=98) who accepted to participate and fulfilled inclusion criteria were randomly allocated to either the intervention or control group by chart number while their TKA was being scheduled in the orthopedic outpatient department (OPD). The researcher was blinded to the randomization in order to prevent the knowledge of the allocated interventions.

Of those 98 patients, 10 individuals withdrew from the study, at different stages, due to different reasons (4 patients had postoperative complications, 4 patients did not want to continue in the study and 2 patients moved to another city). Finally, 44 patients were allocated to the intervention group and 44 patients to the control group.

Baseline testing occurred 6 weeks before the participant's scheduled TKA. All 88 participants were asked to complete the questionnaire package, which consisted of the following: 1) demographic questionnaire, 2) WOMAC score questionnaire, 3) Knee Injury and osteoarthritis Outcome score (KOOS) questionnaire and 4) Short Form-36 Health Survey (SF-36).

After completing the questionnaires, the participants performed the timed 20-meters flat surface walking test, the timed chair stand test and the isometric quadriceps extension assessment to assess the functionally of knee joint (using an isokinetic dynamometer Humac Norm, Computer Sports Medicine Inc., Massachusetts, USA)

The participants again completed the questionnaires and physical testing at the end of the 6-week intervention, as well as at 4 and 12 weeks after their total knee arthroplasty. All outcome measures were blindly assessed in a standardized order at each test by the principal investigator.

Surgical procedures

All patients underwent a TKA, which was implanted with cement with the same standardized preoperative protocol, surgical technique and performed by the same team of 4 experienced orthopaedic surgeons. In all cases, the posterior cruciate ligament was retained, and the operations were performed with use of a tourniquet.

Postoperatively, all patients received the same post-operative rehabilitation protocol at the hospital as a part of the usual care treatment. This program was focused in restoring knee ROM, strength and normal gait. The strength exercises were specially focused on knee extensor strength, starting without external load and progressing by adding a maximum of 2 or 3 kg.

This rehabilitation program was daily performed during four weeks and each session lasted approximately 60 minutes.

Participants

Subjects assigned (N=44) to the intervention group participated in a 6-week preoperative training program, after baseline testing measurements were taken. The intervention group performed supervised progressive resistance training five sessions per week for 6 weeks pre-operatively, and completed a further five sessions per week for 4 weeks postoperatively. On the other hand, subjects assigned to the control group had no physical therapy intervention preoperatively but they followed the same postoperative rehabilitation training program (5 sessions/week for 4 weeks).

Patients of intervention group had a session of preoperative resistance training five days per week for a period of 6 weeks before TKA. Each session was supervised by a physiotherapist specifically trained in progressive resistance training. The duration of each session was approximately 60 minutes. If a participant missed a training session, it was attempted to substitute the session on an alternative day.

Based on 2009 guidelines of the American College of Sports Medicine, progressive resistance training was defined as a concentric/eccentric muscle contraction against a variable or constant external resistance at a constant or variable velocity, where loading is continuously adjusted to ensure progression.

Participants in the intervention group were prescribed a training program that consisted of a 10-minute aerobic warm-up using a treadmill or a stationary bike, followed by a circuit of bilateral lower body exercises (standing calf raise, seated leg press, leg curl, knee extension, knee flexion and hip abduction) in standard strength training machines (Cybex, Owatonna, MN, USA). Three sets of 8 repetitions of each exercise of each exercise were performed with a rest length of 2 minutes between sets and exercises. All exercises started at 60% of their one repetition maximum and increasing gradually by increments of 1-2 kg per week, as tolerated, over the course of the 6-week intervention.

Only in case more repetitions than prescribed could be made, the load was to be increased. All sessions concluded with 2 minutes of stretching exercises of knee extensors, knee flexors and ankle plantar flexors.

Patients in the control group were instructed to "live as usual" for 6 weeks preoperatively. Postoperatively they followed the same progressive training exercise protocol as the intervention group for a period of 4 weeks.

Outcome measures

This study was designed to evaluate the intervention and its effect on a range of clinically related patient self-assessment and performance-based outcome measures. Several studies concluded that the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and the Medical Outcomes Study Short-Form 36 (SF-36) could be recommended as primary measures in treatment studies. A systemic review also showed that overall, regarding patient-reported outcome measures, the KOOS, WOMAC, and SF-36 are the most comprehensively tested tools in this population and are worth considering.

For patient-reported outcome measurement, the Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC) score was available as part of quality control Issues. It was applied in the Greek-language version. All patients completed the questionnaire 6 weeks before the surgical procedure, 2-3 days before TKA and 4 and12 weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years
2. Patients were diagnosed with advanced idiopathic knee OA (according to the radiological criteria of the American College of Rheumatology Guidelines)
3. Patients who were scheduled for unilateral total knee arthroplasty in Orthopedic Clinic of University Hospital of Alexandroupolis

Exclusion Criteria:

* 1) Medical conditions that exercise was contraindicated (i.e cardiopulmonary comorbidities that precluded modest exercise 2) Diseases that affected their functional performance (suffering from neuromuscular or neurodegenerative conditions) 3) Mental diseases 4) Previous hip or knee joint replacement surgery 5) Severe pain on the controlateral limp that would not allow them to follow any pre- or postoperative interventions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change of Quadriceps strength | Baseline testing occurred 6 weeks before the participant's scheduled TKA. The participants again completed the questionnaires and physical testing at the end of the 6-week intervention, as well as at 4 and 12 weeks after their total knee arthroplasty
  All patients performed 3 maximal isometric contractions of the knee extensors at a knee joint angle of 700 (00 = full knee extension) and of the knee flexors at a knee joint angle of 200 with 60 seconds rest in between (Knapik et al., 1983). For further analysis we selected the attempt with the highest peak torque (Nm). The patients performed 6 maximal concentric contractions in full possible range of motion (ROM); the attempt with the highest peak torque was selected for further analysis. Peak torque values were normalized to body weight and reported as Nm/kg
Knee pain | Baseline testing occurred 6 weeks before the participant's scheduled TKA. The participants again completed the questionnaires and physical testing at the end of the 6-week intervention, as well as at 4 and 12 weeks after their total knee arthroplasty
  the Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC) score was applied in the Greek-language version. All patients completed the questionnaire 6 weeks before the surgical procedure, 2-3 days before TKA and 4 and12 weeks postoperatively.
  The WOMAC is a disease-specific, self-administered questionnaire developed to study patients with hip or knee OA and requires about 10-12 minutes to complete. It has a multidimensional scale made up of 24 items grouped into three dimensions: pain (five items), stiffness (two items), and physical function (17 items). The test questions are scored on a scale of 0-4 and the scores for each subscale are summed up, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function.
Daily living activities | Baseline testing occurred 6 weeks before the participant's scheduled TKA. The participants again completed the questionnaires and physical testing at the end of the 6-week intervention, as well as at 4 and 12 weeks after their total knee arthroplasty
  The SF-36 is a valid and reliable instrument for assessing the general health and function of undergoing TKA patients and is a core component of suggested outcome measures for this procedure. The scores of each subscale are normalized to a scale ranging from 0 to 100, with a higher score reflecting a better health status. We used the Greek version of SF-36 Health Survey and we evaluate physical functioning.
  Knee injury and Osteoarthritis Outcome Score (KOOS) is a useful scale in evaluating symptoms and functional status related to knee injury and knee OA. This tool has five subscales, namely pain, symptoms, daily living, sports and recreational activities, and quality of life related to the knee. KOOS has high test-retest reliability.
Knee joint function | Baseline testing occurred 6 weeks before the participant's scheduled TKA. The participants again completed the questionnaires and physical testing at the end of the 6-week intervention, as well as at 4 and 12 weeks after their total knee arthroplasty
  The 20-meter walk test is frequently used in clinical trials and cohort studies involving individuals with OA, as well as in physical therapy. We measured the 20-meter walk course with a measure wheel and we measured how many seconds each patients neede to complete this distance. The investigator stopped timing as soon as the participant's first heel completely crossed the strip of tape.
  Studies reported that the 20-meter walk test has a high test-re-test reliability among patients with end-stage OA awaiting knee replacements Additionally, we used the 30-second chair stand test that involves recording the number of stands a person can complete in 30 seconds. The participant is seated back straight in the middle of a chair without arms (seat height 45 cm).The participant is instructed to fully sit between each stand and encouraged to complete as many full stands as possible within 30 seconds.

IPD SHARING:
Plan to Share IPD: No